CLINICAL TRIAL: NCT05842083
Title: On-site Supportive Communication Training in Doctor-patient Communication: A Randomized, Controlled Trial
Brief Title: On-site Supportive Communication Training in Doctor-patient Communication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vejle Hospital (Other)
Collaborators: Zealand University Hospital (Other); Aalborg University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: On-site SCT
Record Dates: First submitted 2023-04-24; First posted 2023-05-03 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Communication Programs; Communication, Manual; Communication Research; Oncology; Doctor Patient Relation; Job Stress; Burnout; Satisfaction, Patient; Efficacy, Self
MeSH Terms: conditions — Communication; Manual Communication; Neoplasms; Occupational Stress; Burnout, Psychological; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Oncologists will be randomized between the intervention and usual practice.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Each oncologist will have a total of three intervention days with a psychologist sitting in and observing the doctor-patient consultations and subsequently providing feedback.
  Interventions: Behavioral: On-site supportive communication training
- Control (No Intervention): Oncologists in the control group will conduct consultations as usual.

INTERVENTIONS:
Behavioral: On-site supportive communication training — On-site supportive communication training
  Arms: Intervention

SUMMARY:
The goal of this randomized, controlled clinical trial is to test a new concept for communication skills training (on-site supportive communication training (on-site SCT) in cancer care. The study aims to determine the impact of on-site SCT on patients' rating of oncologists' communication abilities.

Oncologists participating in the study will be randomly allocated to the intervention or control group. In the intervention group each doctor will have a total of three intervention days at intervals of 3-4 weeks. On an intervention day, a psychologist will sit in and observe doctor-patient consultations. After the first consultations, 30 minutes are allocated for feedback to the doctor by the psychologist. After the last consultation of the day, 60 minutes are allocated for thorough feedback and establishment of learning goals to focus on until the next intervention day. Doctor's in the control group will conduct communication as usual.

Researchers will compare the control and intervention groups to see if patients' rating of doctors' interpersonal and communication skills increase when the doctors have participated in on-site SCT. The 15-item Communication Assessment Tool (CAT) will be used.

It will also be investigated whether on-site SCT increases the doctors' rating of themselves in relation to communication efficacy and job satisfaction and decrease their experience of burnout.

DETAILED DESCRIPTION:
Oncologists carry a heavy responsibility when delivering information to cancer patients and helping them navigate through decisions about life-altering treatments, survivorship, and end-of-life care. Comprehensive person-centered psychosocial cancer care should be adapted to the individual patient, which is obviously a challenging task (Dilworth, et al. 2014). Individualized and empathic communication, on the other hand, is of substantial importance to patient satisfaction, adherence to treatment, empowerment, and the ability to navigate in the disease trajectory (Gattellari, et al. 2001; Stewart 1995; Vogel, et al. 2009).

The quality of the communication in medical care has been shown to influence health outcomes, as it increases the risk of unnecessary treatment and is linked to insufficient pain relief and higher anxiety levels (Thorne, et al. 2005). Therefore, considerable effort has been dedicated to interventions that may improve the communication skills of healthcare professionals involved in cancer care (Moore, et al. 2018). The primary purpose has been to improve the quality of the doctor-patient-communication including the doctors' interpersonal skills.

Previous papers have suggested direct feedback on observed situations as an ideal method for improving communication skills (Anderson 2012; Burgess, et al. 2020), but to the best of our knowledge, no randomized clinical trials have used patient feedback during on-site training. Studies on communication skills training courses with recorded consultations/role-play have shown significant effect on key communication skills (Fallowfield, et al. 2002) and increased self-efficacy (Ammentorp, et al. 2007). Two studies have demonstrated long-term maintenance of acquired skills (Finset, et al. 2003; Gulbrandsen, et al. 2013). Until now, no effect on burnout has been demonstrated (Bragard, et al. 2010a; Bragard, et al. 2010b).

Clinical supervision and training aims to develop clinical practice and provide a protected space to allow an educational and reflective process to occur. Although there is still no empirical definition of the term supervision (Milne 2007), in 2004 Bernard and Goodyear defined it as "an intervention provided by a more senior member of a profession to a more junior member or members of that same profession"(Bernard 2004). On this premise, psychologists cannot formally supervise doctors and other terms must be used. In this project we therefore use the term "on-site supportive communication training" (on-site SCT) when referring to the intervention given by the psychologists.

Psychologists have a long tradition of working with communication, creating a reflective learning space, making observations and providing feedback. It is therefore highly relevant to use dedicated psychologists to investigate the effect of on-site SCT on the doctors' communication and on their experienced level of self-efficacy, satisfaction and burn-out.

ELIGIBILITY:
Inclusion Criteria:

* Medical doctors
* Employed at the Department of Oncology, Vejle Hospital, University Hospital of Southern Denmark or Aalborg University Hospital, or Zealand University Hospital, Roskilde/Naestved.
* Work in the outpatient clinics at the participating departments

Exclusion Criteria:

* Doctors whose employment contracts will expire during the study and who do not plan to continue working at the department.
* Doctors who are not willing to sign the informed consent form.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Difference in rate of "Excellent" scores on the Communication Assessment Tool between the intervention and the control group. | 6 months
  Patients rate the doctor's communication skills right after the consultation.

SECONDARY OUTCOMES:
Change in oncologists' rating of own communication efficacy according to the "Self-efficacy in Health Communication" tool from before to after on-site communication training. | 6 months
  The Self-efficacy in Health Communication tool consists of 12 questions eliciting the healthcare professionals' perceived self-efficacy in communication with patients using a 10-point scale from "very uncertain" (1) to "very certain" (10).
Change in oncologists' rating of burnout according to part 2 and 3 of the Copenhagen Burnout Inventory tool from before to after on-site communication training. | 6 months
  The reply options in relation to burnout range from 1 (To a very high degree/always), to 5 (To a very low degree/never-almost never)
Change in oncologists' rating of job satisfaction from before to after on-site communication training. | 6 months
  Job satisfaction is measured in Denmark every other year at the nation-wide employee satisfaction survey, which survey offers a large amount of comparable data. Five items directly concerning job satisfaction will be extracted from the survey.

CONTACTS AND LOCATIONS:
Overall Officials: Kerstin Kiis Antonsen, MD, Principal Investigator — University Hospital of Southern Denmark - Vejle Hospital
Locations (1):
- Department of Oncology, University Hospital of Southern Denmark - Vejle Hospital, Vejle, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dilworth S, Higgins I, Parker V, Kelly B, Turner J. Patient and health professional's perceived barriers to the delivery of psychosocial care to adults with cancer: a systematic review. Psychooncology. 2014 Jun;23(6):601-12. doi: 10.1002/pon.3474. Epub 2014 Feb 11. PMID 24519814
- [Background] Gattellari M, Butow PN, Tattersall MH. Sharing decisions in cancer care. Soc Sci Med. 2001 Jun;52(12):1865-78. doi: 10.1016/s0277-9536(00)00303-8. PMID 11352412
- [Background] Stewart MA. Effective physician-patient communication and health outcomes: a review. CMAJ. 1995 May 1;152(9):1423-33. PMID 7728691
- [Background] Vogel BA, Leonhart R, Helmes AW. Communication matters: the impact of communication and participation in decision making on breast cancer patients' depression and quality of life. Patient Educ Couns. 2009 Dec;77(3):391-7. doi: 10.1016/j.pec.2009.09.005. Epub 2009 Oct 1. PMID 19796910
- [Background] Thorne SE, Bultz BD, Baile WF; SCRN Communication Team. Is there a cost to poor communication in cancer care?: a critical review of the literature. Psychooncology. 2005 Oct;14(10):875-84; discussion 885-6. doi: 10.1002/pon.947. PMID 16200515
- [Background] Moore PM, Rivera S, Bravo-Soto GA, Olivares C, Lawrie TA. Communication skills training for healthcare professionals working with people who have cancer. Cochrane Database Syst Rev. 2018 Jul 24;7(7):CD003751. doi: 10.1002/14651858.CD003751.pub4. PMID 30039853
- [Background] Anderson PA. Giving feedback on clinical skills: are we starving our young? J Grad Med Educ. 2012 Jun;4(2):154-8. doi: 10.4300/JGME-D-11-000295.1. PMID 23730434
- [Background] Burgess A, van Diggele C, Roberts C, Mellis C. Feedback in the clinical setting. BMC Med Educ. 2020 Dec 3;20(Suppl 2):460. doi: 10.1186/s12909-020-02280-5. PMID 33272265
- [Background] Fallowfield L, Jenkins V, Farewell V, Saul J, Duffy A, Eves R. Efficacy of a Cancer Research UK communication skills training model for oncologists: a randomised controlled trial. Lancet. 2002 Feb 23;359(9307):650-6. doi: 10.1016/S0140-6736(02)07810-8. PMID 11879860
- [Background] Ammentorp J, Sabroe S, Kofoed PE, Mainz J. The effect of training in communication skills on medical doctors' and nurses' self-efficacy. A randomized controlled trial. Patient Educ Couns. 2007 Jun;66(3):270-7. doi: 10.1016/j.pec.2006.12.012. Epub 2007 Mar 2. PMID 17337337
- [Background] Finset A, Ekeberg O, Eide H, Aspegren K. Long term benefits of communication skills training for cancer doctors. Psychooncology. 2003 Oct-Nov;12(7):686-93. doi: 10.1002/pon.691. PMID 14502593
- [Background] Gulbrandsen P, Jensen BF, Finset A, Blanch-Hartigan D. Long-term effect of communication training on the relationship between physicians' self-efficacy and performance. Patient Educ Couns. 2013 May;91(2):180-5. doi: 10.1016/j.pec.2012.11.015. Epub 2013 Feb 12. PMID 23414658
- [Background] Bragard I, Etienne AM, Merckaert I, Libert Y, Razavi D. Efficacy of a communication and stress management training on medical residents' self-efficacy, stress to communicate and burnout: a randomized controlled study. J Health Psychol. 2010 Oct;15(7):1075-81. doi: 10.1177/1359105310361992. Epub 2010 May 7. PMID 20453053
- [Background] Bragard I, Libert Y, Etienne AM, Merckaert I, Delvaux N, Marchal S, Boniver J, Klastersky J, Reynaert C, Scalliet P, Slachmuylder JL, Razavi D. Insight on variables leading to burnout in cancer physicians. J Cancer Educ. 2010 Mar;25(1):109-15. doi: 10.1007/s13187-009-0026-9. PMID 20082173
- [Background] Milne D. An empirical definition of clinical supervision. Br J Clin Psychol. 2007 Nov;46(Pt 4):437-47. doi: 10.1348/014466507X197415. PMID 17535535
- [Background] Bernard JM, & Goodyear, R. K. Fundamentals of clinical supervision, 2004.
- [Background] Iversen ED, Steinsbekk A, Falbe Vind B, Bangsgaard A, Cold S, Ammentorp J. Translation and cultural adaptation of the Communication Assessment Tool (CAT), developing a Danish and Norwegian version. Int J Qual Health Care. 2019 Dec 31;31(10):748-751. doi: 10.1093/intqhc/mzz020. PMID 31220279
- [Background] Kristensen TS, Borritz M, Villadsen E, Christensen KB. The Copenhagen Burnout Inventory: A new tool for the assessment of burnout. Work & Stress. 2005;19(3):192-207.
- [Background] Axboe MK, Christensen KS, Kofoed PE, Ammentorp J. Development and validation of a self-efficacy questionnaire (SE-12) measuring the clinical communication skills of health care professionals. BMC Med Educ. 2016 Oct 18;16(1):272. doi: 10.1186/s12909-016-0798-7. PMID 27756291
- [Derived] Antonsen KK, Lyhne JD, Johnsen AT, Esser-Naumann S, Poulsen LO, Lund L, Timm S, Jensen LH. Assessing the effect of On-site supportive communication training (On-site SCT) on doctor burnout: a randomized controlled trial. BMC Med Educ. 2025 Jan 23;25(1):112. doi: 10.1186/s12909-025-06710-0. PMID 39849449
- [Derived] Kk A, At J, Lo P, Jd L, L L, S EN, S T, Lh J. Effects of on-site Supportive Communication Training (On-site SCT) on doctor-patient communication in oncology: Study protocol of a randomized, controlled mixed-methods trial. BMC Med Educ. 2024 May 10;24(1):522. doi: 10.1186/s12909-024-05496-x. PMID 38730382